CLINICAL TRIAL: NCT05554458
Title: Implementation and Evaluation of the ChildTaks+ Intervention in the Czech Republic Aimed at COPMI
Brief Title: Implementation and Evaluation of the ChildTaks+ Intervention in the Czech Republic
Acronym: ChildTaks+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Collaborators: UiT The Arctic University of Norway (Other)
Responsible Party: Principal Investigator, Adela Fararova, Investigator, Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ZD-ZDOVA1-019; EEA Norway Grants 2014-2021 (Other Grant/Funding Number: Financial Mechanism Programme Health); GA UK No. 50122 (Other Grant/Funding Number: The Charles University Grant Agency)
Record Dates: First submitted 2022-09-16; First posted 2022-09-26 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Mental Disorder; Mental Health Issue; Parent-Child Relations; Parent-child Problem; Child Mental Disorder; Eating Disorders; Eating Disorders in Adolescence
Keywords: ChildTalks+,COPMI,mental health prevention,eating disorders
MeSH Terms: conditions — Mental Disorders; Neurodevelopmental Disorders; Feeding and Eating Disorders

STUDY DESIGN:
Intervention Model Description: Methods: 66 families with a parent being treated for any mental health disorder and with a child aged 6-18 are recruited by ChildTalks+ therapists, professionals from health, social and educational facilities. Paired allocation into intervention group IG (N = 33) and control group CG (N = 33) is based on the number of risk factors identified in the family. IG and CG complete questionnaires at the baseline assessment (T0), at the post-test assessment (T1), and at the follow-up assessments after 6 months (T2) and 12 months (T3). IG receive the ChildTalks+ intervention within 2 months after T0 and CG after the T3 assessment. Questionnaires are completed by parents and children aged 12/15. Quantitative data will be supplemented with qualitative data from ChildTalks+ therapists working with patients with eating disorders.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Experimental): Paired allocation into intervention group IG (N = 33) and control group CG (N = 33) is based on the number of risk factors identified in the family. IG and CG complete questionnaires at the baseline assessment (T0), at the post-test assessment (T1), and at the follow-up assessments after 6 months (T2) and 12 months (T3).
  Interventions: Behavioral: ChildTaks+ intervention
- Intervention Group (Active Comparator): IG receive the ChildTalks+ intervention within 2 months after T0 and CG after the T3 assessment.
  Interventions: Behavioral: ChildTaks+ intervention

INTERVENTIONS:
Behavioral: ChildTaks+ intervention — The ChildTalks+ Intervention ChildTalks+ is a preventive intervention originally developed in the Netherlands, targeting children up to 18 years of age. It has been implemented in Norway, Italy, and Portugal. It has a clear and well-described theoretical basis focusing on psychoeducation. Its key strategy is to provide feasible and replicable interventions to improve the quality of life of families where parents are affected by a mental disorder.

SUMMARY:
Aims of the study. The aim of this study is to evaluate the effectiveness of the ChildTalks+ intervention and to implement it in education and practice. By delivering the ChildTalks+ intervention, i.e. educating parents about the transgenerational transmission of the disorder, informing them about the impact on their children, strengthening their parenting competencies, supporting communication within the family and informing COPMI about their parents' mental disorder, listening to their needs and providing emotional and social support to the family, the investigators expect the following outcomes: improved family communication, including children's awareness of their parents' mental health problems, improved overall well-being of COPMI, heightened perceptions of parental competence, increased family protective factors, including strengthened social support, sustained over time. Part of the intervention consists of early identification of social-emotional problems in children and referral for further professional help.

The research questions the investigators will focus on are:

* What are the effects of the ChildTalks+ intervention in families where parents have a mental health disorder?
* Is the ChildTalks+ intervention feasible for therapists who treat patients with mental disorder?
* Is the ChildTalks+ intervention feasible in families where one parent has an eating disorder?
* Should the ChildTalks+ intervention be modified for this group of families where parent has an eating disorders?

DETAILED DESCRIPTION:
Background: Children of parents with mental illness - COPMI face a high risk of developing a mental disorder themselves as a result of transgenerational transmission. Without effective interventions, COPMI represent the next generation of psychiatric patients. ChildTalks+ is a preventive intervention, consists of four structured psychoeducational sessions, designed for parents affected by any mental disorder and their children. Its key strategy is to prevent and reduce the risk of mental disorders in COPMI. In this study, given the clinical practice, the investigators include the diagnostic group of patients with eating disorders. The aim of the project, which will run in the Czech Republic, is to implement and evaluate the effectiveness of ChildTalks+ methodology.

Methods: 66 families with a parent being treated for any mental health disorder and with a child aged 6-18 are recruited by ChildTalks+ therapists, professionals from health, social and educational facilities. Paired allocation into intervention group IG (N = 33) and control group CG (N = 33) is based on the number of risk factors identified in the family. IG and CG complete questionnaires at the baseline assessment (T0), at the post-test assessment (T1), and at the follow-up assessments after 6 months (T2) and 12 months (T3). IG receive the ChildTalks+ intervention within 2 months after T0 and CG after the T3 assessment. Questionnaires are completed by parents and children aged 12/15. Quantitative data will be supplemented with qualitative data from ChildTalks+ therapists working with patients with eating disorders.

Discussion: The ChildTalks+ intervention is expected to strengthen parenting competencies and family protective factors, improve family communication, increase awareness of parental mental health issues, and improve the overall well-being of COPMI with long-term sustainable outcomes. The current study will be an important contribution to the international evidence base for the ChildTalks+ program and will help identify key themes in the implementation of other similar preventive interventions.

ELIGIBILITY:
Inclusion Criteria:

* A parent is being treated for any mental disorder (according to DSM-5 or ICD-10 diagnostic criteria).
* A child in the family is between the ages of 6-18.

Exclusion Criteria:

* acute parental substance or alcohol dependence
* acute mental disorder with significant and distressing symptoms, including suicidal tendencies, that require immediate treatment for children or the parent/s
* parental inability to provide consent due to intellectual disability
* and language barrier

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
The health-related Quality of life (KIDSCREEN): children 12 - 18, parents of children 8 - 18 | Up to 14 months
  Improvement in child's overal well-being. Scores are reported as t-values, with higher scores reflecting a higher health-related quality of life.
The Strengths and Difficulties Questionnaire (SDQ) children: 15 - 18,parents of children: 6 - 18 | Up to 14 months
  Improvement in child's overal well-being. Children with higher total difficulty scores show greater psychopathology.
Mental Health Literacy Scale: children 15 - 18 | Up to 14 months
  Increase awareness of parental mental health problems
Eating questionnaire youth version (CHEDE-Q): children 12 - 18 | Up to 14 months
  Detect child behavioral and emotional problems at an early stage
Parents' Evaluations of Developmental Status (PEDS): parents of children 0 - 8 | Up to 14 months
  Detect child behavioral and emotional problems at an early stage
Parenting Sense of Competence (PSOC): parents of children 6 - 18 | Up to 14 months
  Increase in perceiving parental competences. Subscales are rated on a 6-point scale from 1 ("strongly agree") to 6 ("strongly disagree").
Parent-Child Communication Scale (PCCS): children 12 - 18, parents of children 6 - 18 | Up to 14 months
  Open family communication. Responses are coded on a five-point Likert scale ranging from 1 ("almost never") to 5 ("almost always").

CONTACTS AND LOCATIONS:
Overall Officials: Jana Gricová, Master, Study Director — Department of Psychiatry, First Faculty of Medicine, Charles University Prague, Czech Republic
Locations (1):
- Department of Psychiatry First Faculty of Medicine Charles University, Prague, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: Yes
Czech Social Science Data Archive (https://archiv.soc.cas.cz/cz/ CSDA ) is involved in international research structures, i.e. metadata from research will be shared internationally. The data will be stored as FAIR. The metadata from research will be available without restriction.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After June 2024
Access Criteria: Non-commercial usage
URL: https://archiv.soc.cas.cz/cz/

REFERENCES:
- [Derived] Fararova A, Papezova H, Gricova J, Stepankova T, Capek V, Reedtz C, Lauritzen C, van Doesum K. ChildTalks+: a study protocol of a pre-post controlled, paired design study on the use of preventive intervention for children of parents with a mental illness with focus on eating disorders. BMC Psychiatry. 2022 Nov 16;22(1):715. doi: 10.1186/s12888-022-04349-5. PMID 36384579